CLINICAL TRIAL: NCT01860833
Title: EFFECTS OF NSAIDs ON CLINICAL OUTCOMES, SYNOVIAL FLUID CYTOKINE CONCENTRATION AND SIGNAL TRANSDUCTION PATHWAYS IN KNEE OSTEOARTHRITIS
Brief Title: NSAID Treatment in Knee Osteoarthritis
Acronym: NSKO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGOG1
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ibuprofen; Celecoxib; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- diclofenac 75 mg/day (Active Comparator): diclofenac 75 mg once day slow release
  Interventions: Drug: Diclofenac
- diclofenac 150 mg/day (Active Comparator): diclofenac 75 mg bid
  Interventions: Drug: Diclofenac
- ibuprofen 1200 mg/day (Active Comparator): ibuprofen 600 mg bid
  Interventions: Drug: Ibuprofen
- ibuprofen 1800 mg/day (Active Comparator): ibuprofen 600 mg tid
  Interventions: Drug: Ibuprofen
- celecoxib 200 mg/day (Active Comparator): celecoxib 200 mg once day
  Interventions: Drug: Celecoxib
- celecoxib 400 mg/day (Active Comparator): celecoxib 200 mg bid
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Ibuprofen — time of treatment 14 days
  Other Names: Brufen
  Arms: ibuprofen 1200 mg/day; ibuprofen 1800 mg/day
Drug: Celecoxib — time of treatment 14 days
  Other Names: celebrex
  Arms: celecoxib 200 mg/day; celecoxib 400 mg/day
Drug: Diclofenac — time of treatment 14 days
  Other Names: voltaren
  Arms: diclofenac 150 mg/day; diclofenac 75 mg/day

SUMMARY:
Central mechanisms may play a role in pain perception during osteoarthritis (OA).Local inflammation (which involves production of pro-inflammatory cytokines such as interleukin (IL) 4 TNF-alpha, IL-6 and IL-8) is considered to be a major source of pain.

Certain therapies that specifically interfere with the expression or actions of pro-inflammatory cytokines have been explored. NSAIDs have analgesic, antipyretic and anti-inflammatory properties and are extensively prescribed for several musculoskeletal disorders. Indeed, the Osteoarthritis Research Society International (OARSI) recently recommended the use of NSAIDs for management of knee and hip OA in symptomatic patients. These drugs have been shown to influence cytokine metabolism in the synovial fluid of OA patients with satisfactory relief of painful osteoarthritic joints.

The aim of the current study was to explore whether NSAID treatment inhibits TNF-alpha, IL-6, IL-8, and VEGF secretion in the synovial fluid of osteoarthritic joints. In particular, diclofenac, ibuprofen and celecoxib were studied. Under the hypothesis that relationships between proinflammatory cytokines and the clinical status of OA patients are possible, we also evaluated the association between the concentration of these molecules in the osteoarthritic knee synovial fluid and the pain and functional status of patients with OA. The effects of NSAIDS on signal transduction pathways in the synovial membrane were also investigated.

DETAILED DESCRIPTION:
not desired

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the study were:

* older than 50 years and
* had primary knee OA diagnosed according to the clinical and radiological criteria of the American Rheumatism Association.

Further inclusion criteria were:

* clinical signs of joint inflammation (warmth, swelling or effusion) and
* a disease severity grade 2 or 3 according to the Kellgren-Lawrence classification

Exclusion Criteria:

* allergy to NSAIDs,
* progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease),
* history of gastrointestinal ulcer or bleeding,
* a hemoglobin concentration lower than 11.5 g/dL,
* renal diseases (serum creatinine concentration more than 1.2 times the upper limit of the normal range according to the central laboratory definition reference values), or
* liver dysfunction (serum alanine or aspartate transaminase concentrations more than 1.5 times the upper limit of normal range according to the central laboratory definition reference values).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster universities (WOMAC) osteoarthritis index score | 0-14 days
  Womac was used to 77 measure the disease-specific health status of patients before and after the pharmacological treatment.

SECONDARY OUTCOMES:
Naranjo probability scale | 14 days
  The Naranjo probability scale was used to evaluate the development of adverse drug reaction during this study

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gallelli, MD, Principal Investigator — University of Catanzaro
Locations (1):
- Department of Orthopedic and Trauma Surgery, Catanzaro, Italy

REFERENCES:
- [Derived] Gallelli L, Galasso O, Falcone D, Southworth S, Greco M, Ventura V, Romualdi P, Corigliano A, Terracciano R, Savino R, Gulletta E, Gasparini G, De Sarro G. The effects of nonsteroidal anti-inflammatory drugs on clinical outcomes, synovial fluid cytokine concentration and signal transduction pathways in knee osteoarthritis. A randomized open label trial. Osteoarthritis Cartilage. 2013 Sep;21(9):1400-8. doi: 10.1016/j.joca.2013.06.026. PMID 23973155